CLINICAL TRIAL: NCT04864522
Title: Phase I/II Study of Anti-CD3 x Anti-SLAMF7 (Anti-CS-1) Bispecific Antibody Armed Fresh Peripheral Blood Mononuclear Cells (SLAMF7 FPBMC) in Relapsed/Refractory Multiple Myeloma
Brief Title: Phase I/II Study of SLAMF7 FPBMC/CS-1 FPBMC in Relapsed/Refractory Multiple Myeloma
Acronym: MM FPBMC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual due to a crowded field of effective drugs by the time the study opened
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Laahn Foster, Associate Progessor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR200107
Record Dates: First submitted 2021-03-30; First posted 2021-04-29 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Relapsed; Refractory; Fresh Peripheral Blood Mononuclear Cells (FPBMC); Bispecific antibodies
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Intervention Model Description: SLAMF7 FPBMC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SLAMF7 FPBMC (Experimental): Participants will undergo apheresis to collect cells to make SLAMF7 fresh peripheral blood mononuclear cells (FPBMC). These cells will be activated in the lab to fight against multiple myeloma. About 3-4 days after apheresis, participants will start receiving infusions of SLAMF7 FPBMC. Throughout treatment, participants will have blood taken for labs, to check disease status and also to look at immune response. Study treatment will stop if the participant has disease progression.
  Interventions: Drug: SLAMF7 FPBMC

INTERVENTIONS:
Drug: SLAMF7 FPBMC — Participants will receive 8 weekly infusions of SLAMF7 FPBMC, then 8 additional infusions every 2 weeks.
  Other Names: CS-1 FPBMC

SUMMARY:
The purpose of this study is to understand the safety and estimate the efficacy of combining anti-CD3 x anti-SLAMF7 bispecific antibody fresh peripheral blood mononuclear cells (SLAMF7 FPBMC/CS1 FPBMC) for patients with relapsed and/or refractory multiple myeloma. Patients receive 8 weekly doses and then 8 more doses every 2 weeks of SLAMF7 FPBMC by intravenous infusion.

DETAILED DESCRIPTION:
Once subjects are determined eligible, white blood cells (lymphocytes) are collected via leukapheresis procedure. The white blood cells, specifically T cells, are then mixed with two proteins, OKT3 and IL-2, which activate the cells to multiply.

The "activated" T cells are coated with the OKT3 and elotuzumab (an anti-SLAMF7 drug) to produce bispecific fresh peripheral blood mononuclear cells (FPBMC).

About 72 hours after the leukapheresis procedure, SLAMF7 FPBMC infusions will start. After about 8-9 weeks, participants will have another leukapheresis procedure and then receive doses every 2 weeks for 8 more doses. Before, throughout and following SLAMF7 FPBMC, research blood will be collected to better understand immune response. Disease status will be checked regularly during and after study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Must have received ≥ 2 consecutive cycles of treatment which include an immunomodulatory drug, a proteasome inhibitor, and an anti-CD38 monoclonal antibody either used individually or in combination
2. Documented refractory or relapsed myeloma

   * Refractory is defined as progression while on treatment or within 60 days of last treatment
3. Measurable disease based on at least one of the following lab results within 28 days of enrollment

   * Serum IgG, IgA, or IgM M-protein ≥ 1.0 g/dL
   * Urine M-protein ≥ 200 mg excreted in a 24-hr collection sample
   * Involved serum free light chain (FLC) ≥ 100 mg/L provided the FLC ratio is abnormal
4. ECOG Performance Status 0 -2
5. Left Ventricular Ejection Fraction (LVEF) ≥ 45% at rest (MUGA or Echocardiogram)
6. Age ≥ 18 years at the time of consent (Written informed consent and HIPAA authorization for release of personal health information)
7. Females of childbearing potential, and males, must be willing to use an effective method of contraception for the duration of the treatment with study drug plus 90 days (duration of sperm turnover).
8. Adequate cardiac function as defined as:

   * No EKG evidence of acute ischemia
   * No EKG evidence of clinically significant conduction system abnormalities in the opinion of the treating investigator
   * No EKG evidence of > Grade 2 (> 480 ms) QTc prolongation
   * No uncontrolled angina or severe ventricular arrhythmias
   * No clinically significant pericardial disease
   * No history of myocardial infarction (MI) in the last 6 months
   * No Class 3 or higher New York Heart Association Congestive Heart Failure
9. Demonstrate adequate organ function as defined below; all screening labs should be performed within 14 days prior to enrollment.

   * Absolute lymphocyte count ≥ 400/mm3
   * Absolute neutrophil count ≥ 1,000/mm3
   * Platelets ≥ 75,000/mm3
   * Calculated Creatinine Clearance ≥ 30 ml/min
   * Serum total bilirubin ≤ 1.5 x upper limit of normal
   * AST and ALT < 2.5 times normal

Exclusion Criteria:

1. Known hypersensitivity to elotuzumab (Elo)
2. Amyloidosis, Waldenstrom's macroglobulinemia, POEMS syndrome, or known central nervous system (CNS) involvement
3. Receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment.

   * NOTE: Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
4. Active autoimmune disease that has required systemic treatment in the past 2 years before enrollment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
5. Serious non-healing wound, ulcer, bone fracture, major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to enrollment
6. Active liver disease (such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis)
7. HIV positive or known active Hepatitis C (e.g., HCV RNA [qualitative] is detected) or Hepatitis B (e.g. HBsAg reactive) virus
8. Active bleeding or a pathological condition that is associated with a high risk of bleeding (therapeutic anticoagulation is allowed)
9. Has an active infection requiring systemic therapy
10. History of active TB (Bacillus Tuberculosis)
11. Has received a live vaccine within 30 days of enrollment.
12. Anti-myeloma drug therapy (including radiation therapy) ≤ 14 days prior to apheresis
13. History of myocardial infarction (within 6 months of enrollment), stable or unstable angina
14. History of another malignancy within the past 3 years before enrollment. -- Exceptions include:

    * Basal cell carcinoma of the skin or squamous cell carcinoma of the skin,
    * In situ cancers that have undergone potentially curative therapy
15. Prisoners or patients who are incarcerated
16. Patients who are compulsorily detained for treatment of either a psychiatric or physical illness
17. Pregnant or breastfeeding females: Females of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | From time of informed consent through one week following 8th FPBMC infusion
  An adverse event that is considered at least possibly related to SLAMF7 FPBMC and meets at least one of the protocol-defined criteria
Adverse event profile | From time of informed consent through 30 days following last FPBMC infusion
  Severity, frequency, category, seriousness and duration of adverse events

SECONDARY OUTCOMES:
Overall response rate (ORR) | About once a month during study treatment (for about 6 months), then about every 3 months for 3 years or until first progression
  As defined by International Myeloma Working Group (IMWG) response criteria (partial response (PR), very good partial response (VGPR), complete response (CR), stringent CR (sCR)
Minimal Residual Disease (MRD) status | Through first progression of disease (maximum of 3 years from first infusion)
  Assessed by ClonoSeq, only for patients who achieve stringent CR or CR
Overall Survival (OS) | Through 3 years after first FPBMC infusion
  Duration of time from consent through death or 3 years after first FPBMC infusion
Cellular anti-myeloma responses | Multiple timepoints through 12 months after last FPBMC infusion
  IFN-gamma Elispots stimulated by a multiple myeloma cell line
Progression-free survival (PFS) | From informed consent through first progression or 3 years after enrollment
  Duration of time from consent through first progression (or end of follow-up)
Humoral anti-myeloma responses | Multiple timepoints through 12 months after last FPBMC infusion
  Anti-SOX2 IgG antibodies in the serum by specific ELISA
Lymphocyte response following infusions of SLAMF7 FPBMC | Blood samples collected prior to first infusion and then before the second through fifth infusions
  T cell count and count for T cell subpopulations

CONTACTS AND LOCATIONS:
Overall Officials: Laahn Foster, MD, Principal Investigator — University of Virginia
Locations (1):
- Ashley Donihee, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No